CLINICAL TRIAL: NCT07353619
Title: All-on-X (Full-arch Implant-supported Rehabilitation) Stackable Surgical Guides for Maxillary Terminal Dentition: a 2-year Retrospective Analysis
Brief Title: All-on-X Stackable Guides for Maxillary Terminal Dentition
Status: Recruiting | Type: Observational
Sponsor: Menoufia University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, Clinical Professor and principle investigator, Menoufia University
Other Study IDs: ADMNF-002026
Record Dates: First submitted 2026-01-08; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Maxillary All-on-X implant rehabilitation using a fully digital stackable guided surgery workflow with immediate loading. — Patients underwent maxillary full-arch implant rehabilitation using an All-on-X concept performed with a fully digital stackable guided surgery workflow and an immediate loading protocol. Implant placement was planned prosthetically using three-dimensional imaging and digital planning software. Stackable surgical guides were used to facilitate guided bone reduction when indicated and fully guided implant placement.
  Six implants were placed in the maxillary arch under local anesthesia following a standardized surgical protocol. Implants achieving adequate primary stability were immediately restored with a screw-retained provisional fixed prosthesis supported by multi-unit abutments. Patients were followed according to a predefined clinical and radiographic protocol for outcome assessment.
  Other Names: Stackable guided implant surgery

SUMMARY:
This retrospective study will evaluate the clinical performance of maxillary All-on-X(full-arch implant-supported rehabilitation) implant rehabilitation using stackable guided surgery and immediate loading. Implant survival and peri-implant outcomes will be assessed over a 2-year follow-up, with regression analysis will be used to investigate the influence of surgical and prosthetic variables, including basal seating guide design.

DETAILED DESCRIPTION:
This study is a retrospective analysis of data derived from a prospectively maintained clinical database evaluating the clinical performance of maxillary All-on-X implant rehabilitation using a fully digital stackable guided surgery protocol with immediate loading.

Consecutive patients presenting with terminal maxillary dentition were treated with a maxillary All-on-6 implant-supported complete fixed dental prosthesis (ISCFDP) using a prosthetically driven digital workflow. Implant planning was performed using three-dimensional imaging and dedicated implant planning software, allowing for virtual determination of implant number, position, angulation, and depth in relation to the planned prosthesis. Stackable surgical guides were designed and fabricated to allow guided bone reduction when indicated, followed by fully guided implant placement.

All implants were placed under local anesthesia using a standardized surgical protocol. Implants achieving a minimum insertion torque of 35 Ncm were immediately loaded with a screw-retained provisional fixed prosthesis on multi-unit abutments. Occlusal contacts were minimized during the healing phase to reduce functional loading. Patients were followed according to a predefined clinical and radiographic follow-up schedule for a minimum period of two years.

The primary outcome of the study will be implant survival at 6 months after placement. Secondary outcomes will include peri-implant clinical parameters (plaque index, bleeding on probing, and probing depth), marginal bone level changes which will be assessed on standardized periapical radiographs at prosthesis delivery, 1-year, and 2-year follow-up visits, and implant success according to established criteria.

ELIGIBILITY:
Inclusion Criteria:

Adult patients presenting with terminal dentition of the maxillary arch

Rehabilitation with a maxillary All-on-6 implant-supported complete fixed dental prosthesis

Treatment performed using a fully digital stackable guided surgery workflow

Immediate loading with a provisional fixed prosthesis

Availability of complete clinical and radiographic records

Minimum follow-up period of 2 years

Prosthetic design classified as (Fixed prosthesis) FP-1 or FP-2 according to Misch classification

Exclusion Criteria:

Uncontrolled systemic conditions contraindicating implant surgery

History of head and neck radiotherapy

Presence of untreated periodontal or peri-implant infection at the time of surgery

Incomplete or missing clinical or radiographic records

Cases requiring simultaneous bone grafting procedures

Severe maxillary atrophy (Cawood and Howell Class III-V)

Cases requiring FP-3 prosthetic design

Rehabilitation performed without guided surgery or without immediate loading

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with terminal maxillary dentition who underwent rehabilitation with a maxillary All-on-6 implant-supported complete fixed dental prosthesis using a fully digital stackable guided surgery workflow and immediate loading protocol. Patients included had complete clinical and radiographic records available and were followed for a minimum of 2 years. Prosthetic designs were limited to FP-1 or FP-2 according to Misch classification. Patients with uncontrolled systemic conditions, previous head and neck radiotherapy, untreated infections, or requiring simultaneous bone grafting were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Implant Survival Rate | 6 months after implant placement
  Implant survival was defined as the presence of the implant in situ without removal for any reason, including biological or mechanical failure. Survival was assessed clinically and radiographically following implant placement and immediate loading.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed El-Sawy, PhD, Principal Investigator — Menoufia University
Locations (1):
- Faculty of Dentistry, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No
Up on request from the corresponding author